CLINICAL TRIAL: NCT06309329
Title: Randomized Clinical Trial of Parent Training for Veterans With PTSD Symptoms (Strength at Home - Parents RCT)
Brief Title: Strength at Home - Parents RCT
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: VISN 17 Center of Excellence (U.S. Federal Agency)
Collaborators: United States Department of Defense (U.S. Federal Agency); University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Suzannah Creech, Psychologist, VISN 17 Center of Excellence
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1770023-2
Record Dates: First submitted 2024-03-06; First posted 2024-03-13 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Parent-Child Relations

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Strength at Home Parents (Experimental)
  Interventions: Behavioral: Strength at Home Parents
- VA treatment as usual (Active Comparator)
  Interventions: Behavioral: VA treatment as usual

INTERVENTIONS:
Behavioral: Strength at Home Parents — Strength at Home parents is an 8 week trauma-informed and cognitive behavioral tele-health group intervention that aims to improve parenting behaviors and overall parent-child and family functioning among U.S. military Veterans with post-traumatic stress disorder symptoms
  Arms: Strength at Home Parents
Behavioral: VA treatment as usual — VA treatment as usual includes referral to the online resources at veterantraining.va.gov/parenting .
  Arms: VA treatment as usual

SUMMARY:
The goal of this clinical trial is to compare the effect of the Strength at Home Parents intervention to treatment as usual in veterans enrolled for care at VA facilities in VISN 17 on parenting stress and parenting behaviors. The participant population will have elevated PTSD symptoms and parent-child functioning difficulties with an index child between the ages of 3-12. The main question[s]it aims to answer are: • Does Strength at Home Parents improve parenting stress and parenting behaviors in comparison to a no-treatment control condition? • Are gains maintained over time and is there a gender difference in efficacy? Participants will complete 4 online assessments, and if randomized to the intervention group they will complete an 8 week tele-health group program. If randomized to the control group participants will receive a link to the VA parenting resources website and any referrals they would like to have. Researchers will compare Strength at Home Parents to VA treatment as usual see if the group intervention improves parenting stress and behaviors above and beyond the existing resources.

ELIGIBILITY:
Inclusion Criteria:

Eligible participants are veterans enrolled in any VA VISN 17 facility who meet the following inclusion criteria: Current parent to a child between the ages of 3 and 12 (the index child), who resides with the participant or spends at least two days per week with the participant, elevated PTSD symptoms and Parent-child functioning problems.

Exclusion Criteria:

Major neurocognitive disorder likely to impact comprehension of material, including severe TBI .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-03-30 (Actual); Primary Completion 2029-05 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Parenting Stress Index total score | Time 2: 8-16 weeks
  The Parenting Stress Index, 4th edition (PSI) has 120 items scored on a 5-point scale, yielding a parent and child domain scale measuring stress related to parent and child characteristics. These scale scores are combined to yield a total stress score.
Parenting Stress Index total score | Time 3: 16-24 weeks
  The Parenting Stress Index, 4th edition (PSI) has 120 items scored on a 5-point scale, yielding a parent and child domain scale measuring stress related to parent and child characteristics. These scale scores are combined to yield a total stress score.
Parenting Stress Index total score | Time 4: 24-32 weeks
  The Parenting Stress Index, 4th edition (PSI) has 120 items scored on a 5-point scale, yielding a parent and child domain scale measuring stress related to parent and child characteristics. These scale scores are combined to yield a total stress score.

SECONDARY OUTCOMES:
Laxness subscale on the Parenting Scale | Time 2: 8-16 weeks
  The laxness scale is comprised of 11 items measuring permissive, inconsistent discipline
Laxness subscale on the Parenting Scale | Time 3: 16-24 weeks
  The laxness scale is comprised of 11 items measuring permissive, inconsistent discipline
Laxness subscale on the Parenting Scale | Time 4: 24-32 weeks
  The laxness scale is comprised of 11 items measuring permissive, inconsistent discipline
Over reactivity subscale on the Parenting scale | Time 2: 8-16 weeks
  The over reactivity scale (10 items) measures use of emotional, harsh discipline
Over reactivity subscale on the Parenting scale | Time 3: 16-24 weeks
  The over reactivity scale (10 items) measures use of emotional, harsh discipline
Over reactivity subscale on the Parenting scale | Time 4: 24-32 weeks
  The over reactivity scale (10 items) measures use of emotional, harsh discipline

OTHER OUTCOMES:
PTSD Symptom Checklist score | Time 2: 8-16 weeks
  We will measure PTSD with the PTSD Checklist for DSM-5; PCL-5, a 20-item measure on a 5-point scale assessing PTSD symptom severity. Scores range from 0 to 80 with higher scores reflecting increased endorsement of PTSD symptoms.
PTSD Symptom Checklist score | Time 3: 16-24 weeks
  We will measure PTSD with the PTSD Checklist for DSM-5; PCL-5, a 20-item measure on a 5-point scale assessing PTSD symptom severity. Scores range from 0 to 80 with higher scores reflecting increased endorsement of PTSD symptoms.
PTSD Symptom Checklist score | Time 4: 24-32 weeks
  We will measure PTSD with the PTSD Checklist for DSM-5; PCL-5, a 20-item measure on a 5-point scale assessing PTSD symptom severity. Scores range from 0 to 80 with higher scores reflecting increased endorsement of PTSD symptoms.
Quick Inventory of Depressive Symptoms | Time 1: 8-16 weeks
  We will use the Quick Inventory of Depressive Symptoms (QIDS). The QIDS includes 16 items that capture the severity of nine depressive symptoms in the last 7 days.
Quick Inventory of Depressive Symptoms | Time 2: 16-24 weeks
  We will use the Quick Inventory of Depressive Symptoms (QIDS). The QIDS includes 16 items that capture the severity of nine depressive symptoms in the last 7 days.
Quick Inventory of Depressive Symptoms | Time 3: 24-32 weeks
  We will use the Quick Inventory of Depressive Symptoms (QIDS). The QIDS includes 16 items that capture the severity of nine depressive symptoms in the last 7 days.
Total Family Problems Score | Time 2: 8-16 weeks
  The Systematic Clinical Outcome Routine Evaluation (SCORE-15) Index of Family Functioning and Change is a 15-item, self-administered instrument that assesses family problems and includes subscales for family strengths, family difficulties, and family communication. Each item is rated on a 5-point scale where 1 = Describes us: Very well and 5 = Describes us: Not at all. The scores from all individual items can be added together into a total family problem score.
Total Family Problems Score | Time 3: 16-24 weeks
  The Systematic Clinical Outcome Routine Evaluation (SCORE-15) Index of Family Functioning and Change is a 15-item, self-administered instrument that assesses family problems and includes subscales for family strengths, family difficulties, and family communication. Each item is rated on a 5-point scale where 1 = Describes us: Very well and 5 = Describes us: Not at all. The scores from all individual items can be added together into a total family problem score.
Total Family Problems Score | Time 4: 24-32 weeks
  The Systematic Clinical Outcome Routine Evaluation (SCORE-15) Index of Family Functioning and Change is a 15-item, self-administered instrument that assesses family problems and includes subscales for family strengths, family difficulties, and family communication. Each item is rated on a 5-point scale where 1 = Describes us: Very well and 5 = Describes us: Not at all. The scores from all individual items can be added together into a total family problem score.

CONTACTS AND LOCATIONS:
Locations (1):
- Central Texas Veterans Healthcare System, Temple, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
A de-identified copy of study data will be shared on a yearly basis to the National Institute of Mental Health Data Archive registry (e.g., National Institute of Mental Health (NIMH) data archive (NDA)).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: will become available per NDA policy which is subject to change; data will be shared with authorized users upon publication or 1-2 years after the grant end date specified on the first Notice of Award, as defined in the applicable Data Sharing Terms and Conditions.
Access Criteria: Per NIMH NDA in addition Data access requires sponsorship by an Institution on behalf of Recipient